CLINICAL TRIAL: NCT03518645
Title: Optimal Lesion Preparation With Non-compliant Balloons for the Implantation of Bioresorbable Vascular Scaffolds (BVS) -OPRENBIS Study
Brief Title: Optimal Lesion Preparation With Non-compliant Balloons Before Implantation Of Bioresorbable Scaffolds
Acronym: OPreNBiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCRI (Other)
Collaborators: SIS Medical AG (Industry)
Responsible Party: Principal Investigator, Wojciech Zasada, MD, PhD, KCRI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPreNBiS
Record Dates: First submitted 2018-04-20; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease; Angina, Unstable; Angina, Stable
Keywords: Coronary Artery Disease; OPN NC; Angina; Stable; Unstable
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Angina, Stable; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPN strategy (Experimental): The OPN NC Super High Pressure PTCA Balloon will be used as the study device for lesion preparation for BVS Absorb implantation - OPN strategy of lesion preparation. This balloon has a twin layer balloon construction, which allows a very high pressure resistance of 35 bar. The balloon has a 0.016'' lesion entry profile and is available in sizes between 1.5 and 4.5 mm and lengths of 10, 15 and 20 mm.
  Interventions: Device: OPN strategy
- standard strategy (Active Comparator): Predilatation with standard coronary balloon will be performed for lesion preparation for BVS Absorb implantation - standard strategy of lesion preparation.
  Interventions: Device: standard strategy

INTERVENTIONS:
Device: OPN strategy — Predilatation with OPN balloon will be performed as a lesion preparation for BVS Absorb implantation.
  Arms: OPN strategy
Device: standard strategy — Predilatation with standard balloon will be performed as a lesion preparation for BVS Absorb implantation.
  Arms: standard strategy

SUMMARY:
Study aim : To compare a novel strategy of lesion preparation with noncompliant balloons before implantation of BVS.

Hypothesis: Predilatation with non-compliant balloons could facilitate optimal deployment of BVS. By achieving good scaffold apposition a need for post-dilatation could be significantly reduced. This is expected to result in better short- and long-term outcomes.

DETAILED DESCRIPTION:
Study design:

Following pre-dilatation a BVS will be implanted and optical coherence tomography (OCT) will be performed in all patients. After OCT post-dilatation with non-compliant balloons might be performed if this is considered necessary by the treating interventionist. Final OCT will be performed in all patients. 1:1 Randomization of two strategies before the implantation of bioresorbable scaffolds:

* OPN strategy (study group): pre-dilatation with OPN® NC (non-compliant) Super High Pressure PTCA (percutaneous transluminal coronary angioplasty) balloons
* standard strategy (control group): pre-dilatation with a standard (compliant) balloon

Enrolment:

Randomization of 50 patients

* 25 in the OPN strategy (study group)
* 25 in the standard strategy (control group)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Able and willing to give informed consent.
* Willing to comply with specified follow-up evaluations.
* Clinical manifestation of coronary artery disease: stable angina, unstable angina or non-ST-elevation myocardial infarction.
* De novo lesion.
* Angiographic diameter stenosis > 70 % and/or fractional flow reserve <0.80.
* Vessel diameter between 2.5 and 4.0 mm.
* One- or two vessel disease (defined as diameter stenosis > 70 % in vessels with a diameter > 2.5 mm).
* Up to two lesions in one or two vessels can be treated.

Exclusion Criteria:

Patient characteristics

* Pregnant or nursing patient or planned pregnancy in the period up to 1 year following the index procedure.
* Patient with contraindication for 12 months of dual antiplatelet therapy.
* ST-elevation myocardial infarction.
* Any contraindication to the implantation of BVS. Lesion characteristics
* Visible thrombus in coronary angiography
* Chronic total occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Apposition of bioresorbable scaffold immediately after stent implantation following: pre-dilatation with OPN vs. pre-dilatation with standard balloons. | During the index procedure
  Stent apposition will be assessed based on OCT (optical coherence tomography) visualization.

SECONDARY OUTCOMES:
Procedural success defined as successful delivery of the scaffold. | During the index procedure
  The frequency of procedural success will be compared in both study groups.
Need for post-dilatation after initial OCT. | During the index procedure
  The frequency of post-dilatation will be compared in both study groups.
Scaffold apposition after post-dilatation. | During the index procedure
  The scaffold apposition after post-dilatation will be compared based on OCT assessment in both study groups.
Periprocedural complications: dissection, slow- or no flow, dissection requiring additional stent implantation. | During the index procedure
  The frequency of periprocedural complications as dissection, slow-flow, no flow and dissection requiring additional stent implantation will be compared separately in both study group.
Periprocedural myocardial infarction defined as 5x upper reference level elevation of high sensitive Troponin I (in patients with normal pre-procedural Troponin). | During the index procedure
  The frequency of periprocedural myocardial infarction will be compared in both study groups.
In-stent restenosis requiring revascularization within 12 months post-procedure. | 12 months after the index procedure
  The frequency of in-stent restenosis requiring revascularization will be compared in both study groups in 12 months follow-up.
Rate of stent thrombosis according the ARC (academic research consortium) criteria within 12 months post procedure. | 12 months after the index procedure
  The frequency of stent thrombosis will be compared in both study groups in 12 months follow-up.
Death or myocardial infarction within 12 months post procedure. | 12 months after the index procedure
  The frequency of death and myocardial infarction will be compared separately in both study groups in 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, MD, PhD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] Ayton SL, Aslam S, Dattani A, Yeo JL, Gulsin GS, Slomka PJ, Dey D, McCann GP, Singh A. Association of epicardial adipose tissue with markers of cardiac remodelling and clinical outcomes in asymptomatic aortic stenosis. Open Heart. 2026 Feb 9;13(1):e003804. doi: 10.1136/openhrt-2025-003804. PMID 41663151
- [Derived] Cuculi F, Bossard M, Zasada W, Moccetti F, Voskuil M, Wolfrum M, Malinowski KP, Toggweiler S, Kobza R. Performing percutaneous coronary interventions with predilatation using non-compliant balloons at high-pressure versus conventional semi-compliant balloons: insights from two randomised studies using optical coherence tomography. Open Heart. 2020 Jan 23;7(1):e001204. doi: 10.1136/openhrt-2019-001204. eCollection 2020. PMID 32076567